CLINICAL TRIAL: NCT01361789
Title: COX-2 Inhibitor Versus Glucocorticoid Versus Both Combined
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asker & Baerum Hospital (Other)
Responsible Party: Baerum Hospital, Vestre Viken HF
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2004_01927 COX
Record Dates: First submitted 2011-05-26; First posted 2011-05-27 (Estimated); Last update posted 2011-05-27 (Estimated); Status verified 2011-05

CONDITIONS: Rupture of Anterior Cruciate Ligament
Keywords: Arthroscopic reconstruction; Anterior crucial ligament; Coxib; Dexamethasone
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — parecoxib; valdecoxib; Etoricoxib; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- COXIB (Active Comparator): 40 mg parecoxib (Dynastat, Pfizer®) one hour before surgery and 40 mg valdecoxib (prodrug of parecoxib, Bextra, Pfizer®)were given 8 hour after surgery.
  After retraction of parecoxib from the market:
  Etoricoxib (Arcoxia, MSD) 120 mg given one hour before surgery
  Interventions: Drug: parecoxib, valdecoxib, etoricoxib
- Dexamethasone (Active Comparator): dexamethasone 8 mg iv
  Interventions: Drug: Dexamethasone
- COXIB and dexamethasone (Active Comparator): combination of coxib AND dexamethasone
  Interventions: Drug: parecoxib, valdecoxib, parecoxib and dexamethasone

INTERVENTIONS:
Drug: parecoxib, valdecoxib, etoricoxib — 40 mg parecoxib (Dynastat, Pfizer®) one hour before surgery and 40 mg valdecoxib (prodrug of parecoxib, Bextra, Pfizer®)were given 8 hour after surgery.
  After retraction of parecoxib from the market:
  Etoricoxib (Arcoxia, MSD) 120 mg given one hour before surgery
  Arms: COXIB
Drug: Dexamethasone — 8 mg IV
  Arms: Dexamethasone
Drug: parecoxib, valdecoxib, parecoxib and dexamethasone — combination of both drugs
  Arms: COXIB and dexamethasone

SUMMARY:
Recent studies on molar surgery have shown that a combination of a glucocorticoid and NSAID or COX-2 selective inhibitor gives better pain relief than either of the drugs used separately. The investigators group has also shown that adding dexamethasone on top of a regimen of paracetamol, NSAID and local anesthesia resulted in 45% painfree patients at rest after ambulatory breast cancer surgery.

The goal of this study is to test the NSAID + glucocorticoid concept in ACl repair. The investigators want to evaluate whether a selective COX-2 selective inhibitor or a glucocorticoid or a combination of both drugs, as part of a multimodal analgesic regime, can provide improved pain relief and shorter hospital stay in patients undergoing outpatient ACL surgery.

ELIGIBILITY:
Inclusion Criteria:

* Arthroscopic reconstruction of the anterior crucial ligament (ACL)
* At least 18 years old
* ASA I + II

Exclusion Criteria:

* Known renal impairment
* Liver failure and/-or an asthmatic condition
* Pregnancy
* Breast feeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2004-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Postoperative VAS score at rest 24 hours after surgery | 24 hours

SECONDARY OUTCOMES:
Cumulated opioid consumption | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Vegard Dahl, PhD, Principal Investigator — Baerum Hospital; Ulrich J Spreng, MD, Principal Investigator — Baerum Hospital
Locations (1):
- Baerum Hospital, Rud, Norway